CLINICAL TRIAL: NCT02924922
Title: Robot Assisted Partial Nephrectomy (RAPN) in Selective Ischemia Versus Laparoscopic Partial Nephrectomy (LPN) in Total Ischemia: Prospective Randomized Study to Assess Oncological and Functional Outcomes
Brief Title: Assessment of Oncological and Functional Outcomes After Robot Assisted Partial Nephrectomy Versus Laparoscopic Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Principal Investigator, Agostino Mattei, Ass. Prof. Dr. med., Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKNZ 2015-446
Record Dates: First submitted 2016-09-23; First posted 2016-10-05 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Kidney Neoplasms
Keywords: renal cell carcinoma; laparoscopic partial nephrectomy; robot-assisted partial nephrectomy; nephron sparing surgery; warm ischemia time; renal function loss
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic partial nephrectomy (Active Comparator): 1. Inclusion criteria fulfilled:
     * Baseline Abdomen CT/MRI
     * Patient Age, Weight, Height, Co-Medication
     * Informed Consent
     * Baseline renal function (eGFR, renal scintigraphy, sCreatinine, creatinine clearance)
  2. During hospitalization, one day before laparoscopic partial nephrectomy:
     * eGFR
     * sCreatinine
     * Hemoglobin
  3. After surgery:
     * Assessment of eGFR 4 days after operation
     * Hb assessment every 6 H in the first 48 H
     * Assessment of adverse events
     * Histological Results
  4. 6, 12, 24 months after intervention:
     * Creatinine Clearance (only performed at 6 months follow-up)
     * Tc-99m MAG3Dynamic Scintigraphy (only performed at 6 months follow-up)
     * eGFR
     * Assessment of adverse events
     * Assessment of possible recurrence
     * Assesment of kidney volume variation
  Interventions: Procedure: Laparoscopic partial nephrectomy; Device: Conventional laparoscopic instruments; Drug: Mannitol
- Robot assisted partial nephrectomy (Active Comparator): 1. Inclusion criteria fulfilled:
     * Baseline Abdomen CT/MRI
     * Patient Age, Weight, Height, Co-Medication
     * Informed Consent
     * Baseline renal function (eGFR, renal scintigraphy, sCreatinine, creatinine clearance)
  2. During hospitalization, one day before robot assisted partial nephrectomy:
     * eGFR
     * sCreatinine
     * Hemoglobin
  3. After surgery:
     * Assessment of eGFR 4 days after operation
     * Hb assessment every 6 H in the first 48 H
     * Assessment of adverse events
     * Histological Results
  4. 6, 12, 24 months after intervention:
     * Creatinine Clearance (only performed at 6 months follow-up)
     * Tc-99m MAG3Dynamic Scintigraphy (only performed at 6 months follow-up)
     * eGFR
     * Assessment of adverse events
     * Assessment of possible recurrence
     * Assesment of kidney volume variation
  Interventions: Procedure: Robot assisted partial nephrectomy; Device: Da- Vinci Robot and conventional laparoscopic instruments; Drug: Mannitol

INTERVENTIONS:
Procedure: Laparoscopic partial nephrectomy — The renal hilus is identified and both vein and artery are dissected. A laparoscopic ultrasound probe is introduced through a 12 mm port to define the tumor resection margins. A laparoscopic Satinsky clamp is used to induce total kidney ischemia, clamping both vein and artery. Athermal resection of the tumor is performed and titanium clips are used to close interlobar or arcuate arteries encountered during resection. The defect is closed with stitches secured by Hem-o-Lok clips and haemostatic glue. Ischemia is interrupted once renorrhaphy is completed
  Other Names: LPN; Minimally invasive partial nephrectomy
  Arms: Laparoscopic partial nephrectomy
Procedure: Robot assisted partial nephrectomy — The renal hilus is carefully dissected, so that the arterial segmental branches are reached. Tumor resection margins are identified through ultrasound. Drop-in bulldog clamps are used to clamp segmental arterial branches and induce selective ischemia. Indocyanine green 0.2-0.3mg/KG is infused intravenously a few seconds after the selective ischemia is induced. The Firefly near infra-red fluorescence system is used to determine the extent of the ischemic area. The ischemic zone can now be tailored to the tumor by adding or removing bulldog clamps according to the vascular anatomical conditions. Athermal resection of the tumor is performed and titanium clips are used to close interlobar or arcuate arteries encountered during resection. The resection defect is closed with stitches secured by Hem-o-Lok clips and haemostatic glue. Selective ischemia will be interrupted once renorrhaphy is completed
  Other Names: RAPN; Da Vinci; Robot assisted minimally invasive surgery
  Arms: Robot assisted partial nephrectomy
Device: Conventional laparoscopic instruments — Endoscope, Scissor, Needleholder, Forceps, Suction unit, Ports, Tissel, CO2, Sutures, Needles, Scalpel, Ultrasound-Probe, Monitors
  Arms: Laparoscopic partial nephrectomy
Device: Da- Vinci Robot and conventional laparoscopic instruments — Da Vinci Robot, Console, Ports and Instruments; Suction unit, Forceps, Tisseel, Ultrasound Probe, Monitors
  Arms: Robot assisted partial nephrectomy
Drug: Mannitol

SUMMARY:
Currently, partial nephrectomy (PN) is considered as the gold standard treatment modality for small renal masses. In this setting, robot-assisted and conventional laparoscopic approaches are gaining more consensus every day. However, until now, no superiority of one technique over the other has yet been demonstrated, especially on postoperative function recovery.

This study compares oncological and functional outcomes after laparoscopic partial nephrectomy versus robot assisted partial nephrectomy.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) represents 2-3% of all cancers, with the highest incidence in Western countries. Due to increased detection of tumors by ultrasound (US) and computed tomography (CT), the number of incidentally diagnosed RCCs has increased. These tumors are usually smaller and of lower stage. Currently, partial nephrectomy (PN) is considered as the gold standard treatment modality for small renal masses. In this setting, robot-assisted and conventional laparoscopic approaches are gaining more consensus every day. However, until now, no superiority of one technique over the other has yet been demonstrated, especially on postoperative function recovery. This is a single center prospective randomized trial investigating the functional and oncological outcomes of minimally invasive (laparoscopic and robot-assisted) nephron sparing surgery. Patients will be assessed with renal scintigraphy and 24 hours creatinine clearance pre- and postoperatively. Furthermore, duration of the operation, resection and suturing times will be assessed. Renal function recovery is defined as primary endpoint; oncological outcome and positive surgical margin rate are defined as secondary measures. In addition, kidney volume variation will be calculated to describe the amount of healthy tissue preserved in both procedures.The aim of the study is to assess whether robot assisted partial nephrectomy in selective ischemia is superior to laparoscopic partial nephrectomy in global ischemia in terms of functional and oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years
* Organ-confined renal cancer (tumor stage cT1-cT2), assessed by MRI/CT
* Patient qualifies for robotic or laparoscopic partial nephrectomy
* Written informed consent

Exclusion Criteria:

* Renal masses necessitating radical tumor nephrectomy
* Patients with single kidney
* Bilateral kidney cancer when simultaneously operated
* Previous partial nephrectomy
* Renal insufficiency: Chronic Kidney Disease (CKD) stages 4-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change of Scintigraphic Split Renal Function (%) after surgery | Scintigraphic split renal function (%) preoperatively and at 6 months follow up

SECONDARY OUTCOMES:
Duration of Operation | During surgery
Duration of Warm Ischemia | During surgery
Mass Resection Time | During surgery
Suturing Time | During surgery
Amount of Spared Renal Parenchyma | During surgery
Rate of Recurrence | 6 months - 12 months - 24 months
Positive Surgical Margin Rate | During surgery

OTHER OUTCOMES:
Change of Renal Function After Surgery (eGFR) | eGFR assessment preoperatively, first postoperative day and at all follow ups (6, 12, 24 months)
Change of Renal Function After Surgery (sCreatinin) | Serum creatinine preoperatively, first postoperative day and at all follow ups (6, 12, 24 months)
Change of Renal Function After Surgery (24 hour Creatinin Clearance) | 24 hour Creatinin Clearance preoperatively and at 6 months follow up
Change of Hemoglobin after Surgery (Hb) | Preoperatively, 6 hours postoperatively, 12 hours postoperatively, 18 hours postoperatively, 24 hours postoperatively, 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Mattei, Ass. Prof., Principal Investigator — Luzerner Kantonsspital Luzern, Leiter der Klinik für Urologie
Locations (1):
- Klinik für Urologie, Kantonsspital Luzern, Lucerne, Switzerland